CLINICAL TRIAL: NCT06981559
Title: A Clinical Study on the Impact of Hemoperfusion on the Prognosis of Uremic Patients Undergoing Maintenance Hemodialysis
Status: Not yet recruiting | Type: Observational
Sponsor: xujiao chen (Other)
Responsible Party: Sponsor-Investigator, xujiao chen, Professor, Huashan Hospital
Organization: Huashan Hospital (Other)
Other Study IDs: KY2024-1356
Record Dates: First submitted 2025-04-15; First posted 2025-05-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-04

CONDITIONS: Hemodialysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- high-frequency hemoperfusion group: ≥1 session every 2 weeks

SUMMARY:
The goal of this real-world clinical trial study is to evaluate the impact of hemoperfusion on the prognosis of patients with End-Stage Renal Disease (ESRD) undergoing maintenance hemodialysis.

DETAILED DESCRIPTION:
The investigators are planning to conduct a real-world clinical trial study, enrolling patients with maintenance hemodialysis (MHD) from Huashan Hospital. Patients will be divided into two groups based on their hemoperfusion (HP) treatment frequency: high-frequency HP treatment group (≥1 session every 2 weeks) and low-frequency HP treatment group (<1 session every 2 weeks). The investigators will collect baseline demographic data, cardiovascular events, cognitive function status, and nutrition-related clinical indicators for both groups. After a 3-year follow-up, The investigators will reassess these parameters to explore the impact of HP on the prognosis of MHD patients.

ELIGIBILITY:
Inclusion Criteria:

Patients undergoing maintenance hemodialysis for ≥3 months Aged ≥18 years and <85 years; Regular hemodialysis treatment, 3 times per week No residual renal function (urine output <200 mL/d); Written informed consent has been obtained from the participant.

Exclusion Criteria:

Patients with severe cerebrovascular diseases (new-onset cerebral infarction, cerebral hemorrhage) or neurological diseases (autoimmune encephalitis, epilepsy, neurodevelopmental disorders).

Patients with acute severe infections (such as sepsis), severe cardiopulmonary insufficiency (NYHA class IV heart failure, acute exacerbation of COPD), or malignancies.

Patients receiving combined hemodialysis and peritoneal dialysis treatment. Patients with allergic reactions, contraindications, or intolerance to dialysis membrane materials.

Patients with a platelet count <60 × 10^9/L. Other conditions deemed by the investigators as unsuitable for participation in this study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be divided into two groups based on the frequency of hemoperfusion treatments they receive: the high-frequency hemoperfusion group (≥1 session every 2 weeks) and the low-frequency hemoperfusion group (<1 session every 2 weeks).
Sampling Method: Non-Probability Sample
Enrollment: 162 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2028-04-30 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with MCI as assessed by Montreal Cognitive Assessmen | month 12 and month 36
  Montreal Cognitive Assessment: A score of 24 or higher is considered normal, while a score below 24 may indicate mild cognitive impairment(MCI）
Number of participants with cardiovascular events according to ACC/AHA guideline | month 12 and month 36
  Number of participants with cardiovascular events including myocardial infarction, stroke, hospitalization for heart failure, or cardiovascular death
Number of participants with Sarcopenia as assessed by using BIA | month 12 and month 36
  ASMI (kg/m2) will be calculated as ASM(kg)/height 2（m2). ASM will be measured using bioimpedance analysis (BIA)

SECONDARY OUTCOMES:
Toxin removal efficiency | month 12 and month 36
  Decline rate of β2-MG from baseline level
Solute removal efficiency | month 12 and month 36
  spKt/V
Toxin removal efficiency | month 12 and month 36
  Decline rate of IL-6 from baseline level
Toxin removal efficiency | month 12 and month 36
  Decline rate of proteomics and metabolomics from baseline levels
Solute removal efficiency | month 12 and month 36
  URR
Solute removal efficiency | month 12 and month 36
  electrolytes (potassium)
Solute removal efficiency | month 12 and month 36
  electrolytes (sodium)
Solute removal efficiency | month 12 and month 36
  electrolytes (calcium)
Solute removal efficiency | month 12 and month 36
  electrolytes (phosphorus)